CLINICAL TRIAL: NCT02840708
Title: SK-1401 (rhGM-CSF Agent for Inhalation) GM-CSF Inhalation Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Niigata University Medical & Dental Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTU
Record Dates: First submitted 2016-07-13; First posted 2016-07-21 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Alveolar Proteinosis, Autoimmune
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired | interventions — sargramostim

ARMS (3):
- 125mcg (Active Comparator): SK-1401 125mcg single inhalation
  Interventions: Drug: Sargramostim
- 250mcg (Active Comparator): SK-1401 250mcg single inhalation
  Interventions: Drug: Sargramostim
- 500mcg (Active Comparator): SK-1401 500mcg single inhalation
  Interventions: Drug: Sargramostim

INTERVENTIONS:
Drug: Sargramostim

SUMMARY:
Objective: Evaluate Pharmacokinetics and determine the safety of GM-CSF single dose inhalation.

Study Design: Pharmacokinetic open study

ELIGIBILITY:
Inclusion Criteria:

1. Subjects judged to be appropriate for the study by the attending physician
2. can provide signed informed consent.

   aPAP patient must meet the following
3. aPAP patient aged over 20 and below 80 years old (as of the date of registration)
4. aPAP severity is mild or moderate. (not severe)

   Healthy volunteer must meet the following
5. Japanese healthy male subject aged over 20 and below 45 years old (as of the date of registration).
6. BMI (Body mass index) is between 18 and 25.

Exclusion Criteria:

1. WBC of 12,000/mcl or more
2. Fever of 38 degree celsius or more
3. History of malignant disease within recent 5 years (not applied to the treated cases of local basal cell carcinoma)
4. Complication of severe cardiovascular diseases including congestive heart failure, angina pectoris, hemorrhagic tendency, etc.
5. Complication of respiratory diseases such as pulmonary infectious disease(incl. pulmonary tuberculosis), interstitial pneumonitis, lung fibrosis or bronchiectasis, in which the evaluations of safety of GM-CSF therapy are considered to be difficult.
6. History or complication of infectious diseases which require systemic administration of antibiotics, antifungal or antiviral agents within recent 2 weeks.
7. liver dysfunction
8. renal dysfunction
9. Previous experience of severe and unexplained adverse events during aerosol delivery of any kind of medicinal product
10. Positive for HIV-Ab, HBs-Ag, HCV-Ab, STS or TPHA
11. allergic to GM-CSF.
12. addicted to illegal drugs
13. Participation to other clinical trials within 12 weeks before registration.
14. smoking within 5 years
15. cannot follow the procedure defined in this protocol

    aPAP patient must exclude the following
16. Pregnant or possibly pregnant women, lactating women, and women who desire to become pregnant during the study period
17. Patients who have been treated with whole-lung lavage, repeated segmental-lung lavage, GM-CSF or rituximab within 6 months before the start of the study.
18. taking other inhalation.

    Healthy volunteer must exclude the following
19. taking any medicines (incl. OTC).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Serum level of Sargramostim | 0.5,1,2,4,8,12 and 24 hours after inhalation

CONTACTS AND LOCATIONS:
Locations (1):
- Niigata University Med & Dental Hospital, Niigata, Japan